CLINICAL TRIAL: NCT06957886
Title: A Randomized, Controlled Phase III Study of BL-M07D1 Versus Investigator's Choice of Chemotherapy in Patients With HER2-low Recurrent/Metastatic Breast Cancer
Brief Title: A Study of BL-M07D1 Versus Investigator's Choice of Chemotherapy in Patients With HER2-low Recurrent/Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-304
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: HER2-low Breast Cancer
MeSH Terms: interventions — Capecitabine; eribulin; Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-M07D1 (Experimental): Participants receive BL-M07D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1
- investigator's choice of chemotherapy (Active Comparator): Participants receive Capecitabine, Eribulin, Gemcitabine, Paclitaxel, or Albumin paclitaxel for the first cycle. Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Capecitabine, Eribulin, Gemcitabine, Paclitaxel, or Albumin paclitaxel

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: BL-M07D1
Drug: Capecitabine, Eribulin, Gemcitabine, Paclitaxel, or Albumin paclitaxel — Oral administration of Capecitabine. Administration by intravenous infusion of Eribulin, Gemcitabine, Paclitaxel, or Albumin paclitaxel.
  Arms: investigator's choice of chemotherapy

SUMMARY:
This trial is a registered, phase III, randomized, open-label and multicenter study to evaluate the efficacy and safety of BL-M07D1 in patients with unresectable, locally recurrent or metastatic HER2-low breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. Women aged ≥18 years and ≤75 years at the time of written informed consent;
3. Expected survival time ≥12 weeks;
4. Histologically or cytologically confirmed unresectable, locally recurrent or metastatic HER2-low breast cancer;
5. Provide the latest tumor tissues to the central laboratory for HER2 and HR detection;
6. Meet the treatment requirements in the plan;
7. Must have at least one measurable target lesion that meets the RECIST v1.1 definition;
8. ECOG 0 or 1;
9. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
10. Organ function level must meet the requirements;
11. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, serum pregnancy must be negative, and must be non-lactating; All enrolled patients (male or female) should use adequate, highly effective contraception for the entire treatment cycle and for 7 months after completion of treatment.

Exclusion Criteria:

1. Received mitomycin C and nitrosourea chemotherapy within 6 weeks before the first dose, and received surgery or radical radiotherapy within 4 weeks before the first dose;
2. Patients who were not suitable to use the control drugs chosen by the researchers because of intolerance to the chemotherapy drugs of the control group or other contraindications;
3. Previous treatment with anti-HER2 drugs;
4. Prior ADC drug therapy with camptothecin derivative as toxin;
5. The history of severe cardiovascular and cerebrovascular diseases in the past six months was screened;
6. Severe impairment of lung function due to concurrent pulmonary diseases;
7. History of ILD/interstitial pneumonia requiring steroid therapy, current ILD/interstitial pneumonia or suspected ILD/interstitial pneumonia;
8. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
9. Other primary malignancies diagnosed within 5 years before the first dose;
10. Poorly controlled hypertension;
11. Patients with active central nervous system metastases;
12. Patients with a history of severe allergy to any excipients or components of the study drug;
13. History of autologous or allogeneic stem cell transplantation or organ transplantation;
14. Anthracycline-equivalent cumulative dose of adriamycin > 360 mg/m2;
15. Human immunodeficiency virus antibody positive, active hepatitis B virus infection, cirrhosis, or hepatitis C virus infection;
16. Serious infection within 4 weeks before the first dose of study drug; Severe infection requiring antibiotic, antiviral or antifungal control at screening;
17. Patients with massive effusions, or effusions with obvious symptoms, or poorly controlled effusions;
18. Carcinomatous lymphangitis;
19. Was receiving &gt before randomization; 10mg/d prednisone systemic corticosteroids or equivalent anti-inflammatory active drugs or any form of immunosuppressive therapy;
20. The presence of a severe neurological or mental illness;
21. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
22. Intestinal obstruction, Crohn's disease, ulcerative colitis or chronic diarrhea;
23. Subjects who are scheduled to receive live vaccine or receive live vaccine within 28 days before the first dose;
24. Patients with other serious physical or laboratory abnormalities or poor compliance that may increase the risk of participating in the study or interfere with the results of the study, and patients who are considered by the investigators to be unsuitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 566 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BICR is defined as the time between the date subjects were randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Clinical Benefit Rate (CBR) | Up to approximately 24 months
  Clinical benefit ratio (CBR) is defined as the percentage of patients with advanced cancer who achieved complete remission, partial remission, or stable disease for at least 6 months after treatment.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-M07D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan